CLINICAL TRIAL: NCT00000242
Title: Carbamazepine Treatment of Cocaine Dependence
Brief Title: Carbamazepine Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-07761-1; R29DA007761 (NIH); R29-07761-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 1996-07

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: Cocaine; Substance Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The purpose of this study is to compare the efficacy of carbamazepine in treatment of cocaine-dependence in patients with affective disorders.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1992-10-01 (Actual); Primary Completion 1997-01-25 (Actual); Study Completion 1997-01-25 (Actual)

PRIMARY OUTCOMES:
Severity addiction
Amount of drug use
Affective stability
Medication compliance

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Brady, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Brady KT, Sonne S, Randall CL, Adinoff B, Malcolm R. Features of cocaine dependence with concurrent alcohol abuse. Drug Alcohol Depend. 1995 Jul;39(1):69-71. doi: 10.1016/0376-8716(95)01128-l. PMID 7587977